CLINICAL TRIAL: NCT07038629
Title: Concurrent Chemoradiation Plus Iparomlimab Consolidation Therapy for Older Patients With Inoperable Locally Advanced Esophageal Squamous Cell Carcinoma: A Single-arm Phase II Clinical Study
Brief Title: Chemoradiation Plus Iparomlimab Consolidation in Older With ESCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Shanxi Province Cancer Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20250418
Record Dates: First submitted 2025-05-21; First posted 2025-06-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Cancer
Keywords: Old Age; Esophageal Cancer; Iparomlimab; Chemoradiation
MeSH Terms: conditions — Esophageal Neoplasms | interventions — S 1 (combination); Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemoradiation Plus Iparomlimab Consolidation (Experimental): S1 + Radiotherapy+ Iparomlimab Consolidation:
  Chemotherapy: S1 PO, 40~60mg，BID（d1-14，d22-35，two cycles); Radiation: Concurrent Radiation, 1.8Gy/f, 28f; Iparomlimab Consolidation: Iparomlimab IV infusion, 5mg/kg, q3w (Started within 8 weeks of completion of radiation)
  Interventions: Drug: S1; Drug: Iparomlimab; Radiation: Radiation

INTERVENTIONS:
Drug: S1 — PO, 40~60mg，BID（d1-14，d22-35，two cycles)
Drug: Iparomlimab — IV infusion, 5mg/kg, q3w (Started within 8 weeks of completion of radiation)
Radiation: Radiation — Concurrent Radiation, 1.8Gy/f, 28f;

SUMMARY:
This study was conducted in elderly (≥70 years old) patients with locally advanced esophageal squamous cell carcinoma (ESCC). Aim to evaluate the efficacy and safety of Iparomlimab consolidation therapy following concurrent chemoradiation with S-1 in elderly patients with unresectable locally advanced ESCC.

Concurrent chemoradiation is the standard treatment for elderly esophageal cancer. However, the overall prognosis of patients still needs to be further improved. The emergence of immune checkpoint inhibitors has brought new hope for patients with ESCC. Iparomlimab can target both PD-1 and CTLA-4 immune inhibitory pathways simultaneously. Studies have shown that it can significantly improve the prognosis in the treatment of ESCC and has good tolerability. In elderly patients with ESCC, concurrent chemoradiation may potentially carry the risk of low treatment completion rate and significant toxicity. Therefore, this study aims to explore the efficacy and safety of Iparomlimab consolidation therapy following concurrent chemoradiotherapy in elderly patients with unresectable locally advanced ESCC.

In the study, the investigators plan to enroll 52 elderly subjects with locally advanced ESCC. After receiving radiotherapy combined with the S-1 regimen, patients will enter the screening period. The enrolled patients will receive Iparomlimab consolidation therapy for 1 year. The treatment efficacy and safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteered to participate, cooperated with follow-up visits;
2. Aged ≥ 70 years, both male and female;
3. Histologically confirmed cT1N2-3M0 or cT2-4bN0-3M0 or cT1-4bN0-3M1(supraclavicular lymph node metastasis) locally advanced ESCC (8th AJCC );
4. Presence of measurable and/or non-measurable lesions as defined by Japanese Classification of Esophageal Cancer (12th Edition);
5. Initial treatment: definitive concurrent chemoradiotherapy (radiotherapy: total dose 50.4 Gy, delivered in 28 fractions, 1.8 Gy per fraction, 5 times per week; chemotherapy: S-1: 40-60mg, BID, d1-14, d22-35, for a total of 2 cycles).

   1. Radiotherapy: completed ≥ 25 fractions or more (i.e., radiotherapy dose ≥ 45 Gy), S-1chemotherapy: completed at least one cycle (d1-14);
   2. Haven't received any previous systemic anti-tumor therapy before radiotherapy (including but not limited to systemic chemotherapy, radiotherapy, molecularly targeted drug therapy, immunotherapy, biologic therapy, topical therapy and other investigational treatment drugs);
6. ECOG performance status 0 or 1;
7. Provide fresh or archived tumour tissue samples within 6 months (fresh samples preferred) for biomarker analysis (e.g.PD-L1). Sample types are formalin-fixed, paraffin-embedded [FFPE] tumour tissue blocks or at least 5 unstained, 3-5 μm thick FFPE tumour tissue sections;
8. Expected survival of ≥ 3 months.
9. The function of major organs meets the following requirements:

   1. Absolute neutrophil count (ANC) ≥ 1.5×10^9/L;
   2. Platelets ≥ 100×10^9/L;
   3. Hemoglobin ≥ 9g/dL;
   4. Serum albumin ≥ 2.8g/dL;
   5. Total bilirubin ≤ 1.5 × ULN, ALT, AST and/or ALP ≤ 2.5 × ULN;
   6. Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 60mL/min;
   7. International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5× ULN (subjects on stable doses of anticoagulation therapy, such as low molecular weight heparin or warfarin, and with INR within the expected therapeutic range of the anticoagulant can be screened);
10. Documented informed consent.

Exclusion Criteria:

1. Surgery for esophageal cancer;
2. Esophageal fistulae due to infiltration of the primary tumor；
3. Risk of gastrointestinal bleeding, esophageal fistula or esophageal perforation;
4. Patients who developed ≥ grade 2 pneumonia after concurrent chemoradiotherapy with S-1;
5. Poor nutritional status, weight loss of ≥10% in the previous 2 months, with no significant improvement after nutritional intervention;
6. Major surgery or severe trauma within 4 weeks prior to first use of study drug;
7. Uncontrollable pleural effusion, pericardial effusion, or ascites that requires repeated drainage;
8. Received or receiving any of the following treatments in the past:

   1. Anti-PD-1 or anti-PD-L1 antibody therapy, chemotherapy, radiotherapy or targeted therapy;
   2. Participation in a study of an investigational agent or device within 4 weeks before the first dose of study treatment;
   3. Systemic treatment with corticosteroids (>10 mg prednisone equivalent dose per day) or other immunosuppressive agents is required for 2 weeks before the first dose of study treatment(except for the use of corticosteroids for local inflammation of the esophagus and for the prevention of allergy and nausea and vomiting). Other special circumstances need to be communicated to the sponsor. Inhaled or topical steroids and adrenocorticotropic hormone replacement at doses >10mg/day prednisone efficacy dose are permitted if the patient does not have active autoimmune disease;
   4. Received an anti-tumour vaccine or received a live vaccine within 4 weeks before the first dose of study treatment;
9. Any active autoimmune disease or history of autoimmune disease (e.g., interstitial pneumonitis, uveitis, enteritis, hepatitis, pituitary gland inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism); Except for patients with vitiligo or those who had asthma or allergies in childhood but did not need any intervention as adults; patients with autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone and type I diabetes mellitus treated with stable doses of insulin may be included;
10. Diagnosis of immunodeficiency, including positive HIV test, other acquired/congenital immunodeficiency diseases, organ transplantation and allogeneic bone marrow transplantation;
11. Diagnosis of uncontrolled cardiac clinical symptoms or disease such as: a. NYHA II or above heart failure; b. unstable angina; c. myocardial infarction within 1 year; d. clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
12. Severe infections (CTCAE > grade 2), such as severe pneumonia requiring hospitalisation, bacteraemia, infectious co-morbidities, etc., within 4 weeks before the first use of study treatment; Baseline chest imaging suggestive of active lung inflammation, signs and symptoms of infection requiring oral or intravenous antibiotic treatment within 2 weeks before the first use of study treatment, except for prophylactic antibiotic use;
13. History of interstitial lung disease or non-infectious pneumonia, or pulmonary insufficiency ≥ grade 3 as confirmed by pulmonary function tests;
14. Active tuberculosis infection detected by history or CT examination, or history of active tuberculosis infection within 1 year before enrollment or more than 1 year previously without regular treatment;
15. Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (hepatitis C antibody positive and HCV-RNA above the lower limit of detection);
16. Presence of abnormal sodium, potassium, and calcium laboratory test values greater than grade 1 within 2 weeks prior to randomisation that do not improve with treatment;
17. Known hypersensitivity to large protein preparations, or to any of the components of tirilizumab, or anaphylaxis, hypersensitivity, or contraindication to paclitaxel or cisplatin or to any of the components used within their preparations;
18. Previously diagnosed with any other malignancy before the first use of the investigational drug, except for malignancies with low risk of metastasis and death (5-year survival rate>90%), such as adequately treated basal cell or squamous cell skin cancer or cervical carcinoma in situ.
19. As judged by the investigator, the subject has other factors that may lead to forced termination of the study midway.

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 2 years
  progression-free survival

SECONDARY OUTCOMES:
OS | up to 2 years
  overall survival
ORR | up to 2 years
  overall response rate
DoR | up to 2 years
  Duration of Response
AEs | up to 2 years
  Adverse Events
QoL | up to 2 years
  Quality of Life (QoL) score
CGA | up to 2 years
  Comprehensive Geriatric Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Wencheng Zhang, M.D., Principal Investigator — Tianjin Cancer Hospital
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No